CLINICAL TRIAL: NCT00051272
Title: A Multicenter, Double-blind Randomized Placebo-controlled Comparison of the Effects on Sexual Functioning of Extended-release Bupropion Hydrochloride (300-450mg) and Escitalopram (10-20mg) in Outpatients With Moderate to Severe Major Depression Over an Eight-Week Treatment Period
Brief Title: Effects Of Antidepressants On Sexual Functioning In Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130927
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: depression, sexual dysfunction, orgasm disorder, MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Extended-release Bupropion Hydrochloride

SUMMARY:
This study will evaluate the effects of two antidepression medications on sexual functioning.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder (MDD) with current duration lasting 12 weeks but no greater than 2 years.
* Subjects must engage in sexual activity that leads to orgasm at least once every two weeks.
* Subject must have normal orgasmic function and be willing to discuss with investigator.

Exclusion Criteria:

* Subjects that have arousal or orgasm dysfunction.
* Has previously failed to respond to two adequate trials of antidepressants in past 2 years.
* Subject has other unstable medical disorders.
* Subject has a positive urine test for illicit drug use at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2003-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with orgasm dysfunction. Change from baseline in HAMD-17 total score.

SECONDARY OUTCOMES:
Percent of subjects in remission, HAMD-17. Changes in Sexual functioning Questionnaire. CGI-I and CGI-S. Percent of responders, HAMD-17.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Middletown, Connecticut
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Braintree, Massachusetts
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Yakima, Washington